CLINICAL TRIAL: NCT05746507
Title: Pilot Feasibility of Night Respite Care for Postpartum Mothers With Substance Use Disorder in Residential Treatment Programs
Brief Title: Night Respite for Postpartum Mothers With SUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Davida M. Schiff, MD, Assistant Professor of Pediatrics, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P001377; K23DA048169 (NIH)
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder; Maternal Drugs Affecting Fetus; Postpartum Mood Disturbance; Sleep Disorder; Neonatal Opioid Withdrawal
MeSH Terms: conditions — Opioid-Related Disorders; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Overnight infant respite care provided approximately 3 nights per week for 6 weeks (18 nights total) lasting eight hours per night. Overnight respite care will last for eight hours, with one hour reserved to provide teaching about infant-specific temperament and cues.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Night Respite Care (Experimental): 18 overnight night respite care sessions over six weeks with parental skills provided through teachable moments before and after respite care supports
  Interventions: Behavioral: Night Respite Care

INTERVENTIONS:
Behavioral: Night Respite Care — (see description above)

SUMMARY:
This single arm pilot feasibility study will evaluate the implementation of overnight infant respite care and parenting skills to mothers with substance use disorders in the early postpartum period residing in residential substance use disorder treatment programs.

DETAILED DESCRIPTION:
This single arm pilot feasibility study will evaluate the implementation of overnight infant respite care provided approximately 3 nights per week for 6 weeks (18 nights total) to each of 20 - 25 mothers with substance use disorders in the early postpartum period residing in residential substance use disorder treatment programs. Overnight respite care will last for eight hours, with one hour reserved each morning to provide teaching about infant-specific temperament and cues. The program is a unique public/private/academic partnership with the Massachusetts Department of Children and Families (DCF), Boston Baby Nurse and Nanny (BBNN), two residential treatment programs, and Massachusetts General Hospital.

Partnering with BBNN, Newborn Care Experts interested in providing respite care to families impacted by SUD will be paired with postpartum families residing in two residential treatment programs in the Boston area. New Day in Somerville, MA and Entre Familia in Mattapan, MA will partner with MGH to recruit individuals to complete a screening and baseline intake, receive night respite care, and complete a follow up study visit at the completion of the intervention and at 3 months post intervention.

This study will use mixed methods to understand the feasibility and acceptability of the pilot intervention including experiences of this pilot program through the perspectives of program participants, respite care givers, residential treatment overnight staff, and study staff. Respite caregivers and residential treatment program staff will be invited to participate in interviews after each dyad receives their allotted hours of respite care to reflect on this program participant's specific experience.

BBNN, DCF, and residential treatment program leadership staff, will be invited to participate a focus group once at the completion of the study to understand the feasibility, acceptability, and implementation of this program through the lens of their organizations. They will also be invited to take a short survey aimed at assessing their perception of the intervention's appropriateness and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Caring for an infant under 12 months of age.
* Being the primary caretaker for their infant.
* Having a DSM-5 diagnosis of a substance use disorder.
* Currently residing in a participating residential treatment program or private home setting
* English-speaking or Spanish-speakers with limited English proficiency

Exclusion Criteria:

* Having an untreated serious mental health illness.
* Having an untreated substance use disorder or existing concerns that this person is actively using substances.
* Having a history of prior violence or intimate partner violence in the home.
* Provider concern regarding instability or lack of information about home safety.
* Not actively parenting an infant under 12 months of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female-identifying individuals living in residential treatment programs
Enrollment: 41 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Recruitment and Enrollment | Through study completion up to 3 months
  Total number of individuals approached, consented, and enrolled in the study
Study Feasibility | Through three months following intervention period
  Count of total number individuals completing intervention and retained through study follow up
Study Acceptability | Through three months following intervention period
  Feedback in semi-structured interviews with participants and key stakeholders

SECONDARY OUTCOMES:
Maternal sleep quantity | Through three months following intervention
  Measurement of total nightly sleep using actigraphy device
Ability to fall asleep | Through three months following intervention
  Insomnia Sleep Index (Measured on a scale of 0-28)
Sleep quality | Through three months following intervention
  Single Item Sleep Quality Scale;
Postpartum Sleep Quality | Through three months following intervention
  Postpartum Sleep Quality Scale
Maternal mental health - Depression | Through three months following intervention
  Patient Health Questionnaire-8
Maternal mental health - Anxiety | Through three months following intervention
  General Anxiety Disorder-7
Medication for Addiction Treatment Retention | Through three months following intervention
  Continuation of medication for addiction treatment
Substance use treatment retention | Through three months following intervention
  Retention in residential treatment program
Recovery Capitol | Through three months following intervention
  Brief Assessment of Recovery Capitol (BARC-10)
Parental stress | Through three months following intervention
  Parenting Stress Index
Parental bonding | Through three months following intervention
  Postpartum Bonding Questionnaire;
Parental self-efficacy | Through three months following intervention
  Perceived Parenting Self-Efficacy Questionnaire
Social Support | Through three months following intervention
  Postpartum Social Support Scale
Unnecessary unscheduled healthcare utilization | Through three months following intervention
  ED and Urgent care visits attended
Filings for child abuse/neglect | Through three months following intervention
  51A-filings for child abuse or neglect to MA DCF

CONTACTS AND LOCATIONS:
Overall Officials: Davida M Schiff, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Entre Familia Residential Treatment Program, Mattapan, Massachusetts
  - New Day Residential Treatment Program, Somerville, Massachusetts

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT05746507/ICF_000.pdf